CLINICAL TRIAL: NCT01704560
Title: IMPROVING MEASUREMENT OF PARENTS' UNDERSTANDING OF RESEARCH PERMISSION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Carl D'Angio, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 39377
Record Dates: First submitted 2012-10-04; First posted 2012-10-11 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Improve Parent Understanding of Research Permission

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coversheet to Informed Consent (Experimental): Coversheet attached to Informed Consent.
  Interventions: Other: Coversheet to Informed Consent
- No Coversheet (No Intervention): Standard, full permission form, without the coversheet.

INTERVENTIONS:
Other: Coversheet to Informed Consent — The intervention is a one page cover sheet to be affixed to the front of the standard permission form for the trial for which permission is being sought (attached to application). The form will identify the study as research and contain sections that include investigator contact information, the purpose of the study, a brief description of the study procedures, the alternatives, the voluntary nature, the risks, the potential benefits, a discussion of privacy and confidentiality, the costs and the payments. Each topic will also contain a reference to the page in the consent containing the full description of the topic. The form is designed to have a reading level no higher than 6th to 8th grade. Parents will also receive the full permission form, and all required signatures will still be collected on the permission form.
  Arms: Coversheet to Informed Consent

SUMMARY:
Well-informed potential subjects are presumably better able to make autonomous decisions about the risks and benefits of participating in a research study than those in possession of less information. In actuality, prior research into consent understanding suggests that longer forms offering exhaustive information may inhibit rather than promote understanding. Moreover, technical wording in tools used to measure parent understanding of research permission may also lead to inhibition of understanding. This study will test the hypothesis that, among parents of potential subjects for greater-than-minimal-risk research, two modified and simplified subset of questions from the Deaconess Informed Consent Comprehension Test (DICCT), one oral and open-ended and one written and multiple choice, will increase subject understanding of the nature and risks of the research. The study will enroll the parents of 40 potential neonatal research subjects with an interim analysis of data at 20 subjects. Subjects will review a sham research permission form and will be randomized 1:1 to complete one of the two modified comprehension tests in addition to the DICCT (gold-standard) test. Parents will be given an open-ended survey after the tests in order to qualitatively describe their opinions of each test. A subset of parents who have received the written form will also undergo a cognitive interview about the form. A similar subset will also be given an open-ended survey about a proposed permission form cover sheet. The primary outcome will be the correlation of scores between the DICCT and modified comprehension tests, following the sham informed consent process.

ELIGIBILITY:
Inclusion Criteria:

* Parents of potential subjects eligible for a NICHD Neonatal Research Network (NRN) interventional trial ("Hydrocortisone/Extubation") or greater-than-minimal risk observational trial ("PROP")
* Permission being sought for a qualifying study
* English speaking

Exclusion Criteria:

* Permission has not been previously sought for another qualifying study
* Illiteracy (unable to read simple forms)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03-30 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
DICCT Questionnaire | Within 2 weeks after being approached for participation.
  Score on the post-permission DICCT questionnaire. The DICCT is scored on a 28 point scale, with each of 14 parameters being scored as 0 = incorrect, 1 = partially correct, 2 = correct. The DICCT, in addition to being previously validated, has other advantages. It contains questions that are not directly addressed in the cover sheet, but addressed in the full permission form, such as compensation for injury. These items will serve as valuable internal controls. The DICCT is easily adaptable to written answers, which makes it ideal for further modification in future studies.
  The DICCT will be administered during a structured interview, without a time limit. The parent will be allowed to refer to the permission form to answer the questions.

CONTACTS AND LOCATIONS:
Overall Officials: Carl T D'Angio, MD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - Ann Marie Scorsone, Rochester, New York

REFERENCES:
- [Derived] D'Angio CT, Wang H, Hunn JE, Pryhuber GS, Chess PR, Lakshminrusimha S. Permission form synopses to improve parents' understanding of research: a randomized trial. J Perinatol. 2017 Jun;37(6):735-739. doi: 10.1038/jp.2017.26. Epub 2017 Mar 30. PMID 28358380